CLINICAL TRIAL: NCT00730808
Title: Efficacy and Tolerability of a Preoperative Oral Nutritional Supplement (PreOP Booster) vs. Placebo in Surgical Patients (Pilot Study)
Brief Title: Effectiveness and Tolerability of an Oral Nutritional Supplement (PreOP Booster) Given Before Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Dr. Steffen Benzing, Kabi Innovation Centre, Fresenius Kabi Deutschland GmbH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N-POB-04-NL
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2010-05-19 (Estimated); Status verified 2010-05

CONDITIONS: Rectal Tumors
Keywords: Enteral nutritional regimen prior to surgery
MeSH Terms: conditions — Rectal Neoplasms | interventions — Food

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Test (Experimental): Oral nutritional supplement: assignment according to consecutive random numbers.
  Interventions: Dietary Supplement: PreOP Booster (food for special medical purposes)
- Control (Placebo Comparator): Assignment according to consecutive random numbers.
  Interventions: Dietary Supplement: PreOP Booster (food for special medical purposes)

INTERVENTIONS:
Dietary Supplement: PreOP Booster (food for special medical purposes) — 3x1 dosage is given prior to surgery: 2x1 the day prior to surgery; 1x1 3-4h prior to initiation of anaesthesia;

SUMMARY:
The aim of this pilot study is to investigate effectiveness, tolerability and safety of an oral nutritional supplement (PreOP Booster), given to rectal tumour patients prior to low anterior resection.

ELIGIBILITY:
Inclusion Criteria:

* rectal tumour with indication for elective low anterior resection (open surgery, not laparoscopic surgery) or abdominoperineal resection (APR)
* preoperative radiotherapy (5x5 Gy) or chemoradiation
* loop ileostoma or colostoma;

Exclusion Criteria:

* severe malnutrition
* severe renal insufficiency
* diabetes mellitus I or II
* concomitant thyroid medication
* corticosteroids
* diuretic medication and antihypertensive medication
* known or suspected allergy to any component of the investigational product(s)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Immunoinflammatory parameters | on day -2, -1, 1, 2, 3, 5, and 7
Antioxidant / oxidant parameters | on day -2, 1, 3, 5, and 7
Ischemia / reperfusion injury parameters | on day -2, 1, 3, 5, and 7

SECONDARY OUTCOMES:
pre-and postoperative discomfort (well-being) | on day -1, and 0
hand grip strength | on day -2, 1, 2, 3, 5, and 7
GI tolerance | on day -1, 0, 1, 2, and 7
Safety | on day -1, 0, 1, 2, 3, 5, and 7

CONTACTS AND LOCATIONS:
Overall Officials: Paul A.M. van Leeuwen, Prof., Study Chair — University Hospital Amsterdam; The Netherlands
Locations (1):
- Medical Center Alkmaar, Alkmaar, Netherlands